CLINICAL TRIAL: NCT04258111
Title: An Open-label, Multicenter, Phase 2 Study of IBI310 in Combination with Sintilimab in Patients with DNA Mismatch Repair Deficient (dMMR) /microsatellite Instability High (MSI-H) Locally-advanced or Metastatic Colorectal Cancer
Brief Title: IBI310 in Combination with Sintilimab in Patients with DNA Mismatch Repair Deficient (dMMR)/microsatellite Instability High (MSI-H) Locally-advanced or Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After careful consideration, our company has decided to revise the overall development strategy for IBI310 and discontinue further registration research for this project. Consequently, the ongoing screening process will be terminated, and this decisi
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI310D201
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IBI310 + Sintilimab (Experimental)
  Interventions: Biological: IBI310 (anti-CTLA-4 antibody); Biological: Sintilimab(anti-PD-1 antibody)

INTERVENTIONS:
Biological: IBI310 (anti-CTLA-4 antibody) — Specified dose on specified days
Biological: Sintilimab(anti-PD-1 antibody) — Specified dose on specified days

SUMMARY:
The main purpose of this study is to assess the efficacy and safety of IBI310 in combination with sintilimab in patients with Microsatellite Instability High (MSI-H) or Mismatch Repair Deficient (dMMR) locally advance or metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal adenocarcinoma
2. Imaging confirmed locally-advanced or metastatic colorectal cancer
3. Measurable disease by CT or MRI
4. MSI-H confirmed by central lab
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1

Exclusion Criteria:

1. Prior treatment with an anti-Programmed Death Receptor (PD)-1, anti-PD-L1, anti-PD-L2, anti-Cytotoxic T-Cell Lymphoma-4 Antigen (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
2. Subjects with active,known or suspected autoimmune disease
3. Subjects with a history of primary immune deficiency
4. Subjects with severe infectious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
ORR | Up to 3 years
  Objective Response Rate (ORR) in all MSI-H CRC patients as determined by independent review committee

SECONDARY OUTCOMES:
ORR in all MSI-H CRC patients based on investigator assessment. | Up to 3 years
Progression-Free Survival (PFS) both by investigator and IRC | Up to 3 years
Disease Control Rate (DCR) both by investigator and IRC | Up to 3 years
Duration of Response (DoR) both by investigator and IRC | Up to 3 years
Time To Response (TTR) both by investigator and IRC | Up to 3 years
Overall Survival | Up to 3 years
Incidence of adverse events (AE) | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing cancer hospital, Beijing, China